CLINICAL TRIAL: NCT04725643
Title: Keep Contraceptive Arm Long Acting-iMplant (CALM) and Carry On
Acronym: CALM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sheila Mody, Associate Professor, University of California, San Diego
Other Study IDs: 201908
Record Dates: First submitted 2020-12-16; First posted 2021-01-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Contraception; Contraceptive Usage; Family Planning
Keywords: Nexplanon, Contraceptive implant
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Implant Group: Adults who are choosing to get a replacement Nexplanon and agree to track and report their bleeding patterns for one month before replacement and 3 months after.
  Interventions: Device: Track bleeding patterns before and after implant

INTERVENTIONS:
Device: Track bleeding patterns before and after implant — Participants will report if they had bleeding and the amount based on the Pictorial Blood Assessment Chart. Participants will also complete weekly surveys regarding their satisfaction with their bleeding. We will also ask participants to complete a survey regarding their satisfaction with their bleeding at end of month 2 and at the end of month 3 after replacement of their contraceptive implant.

SUMMARY:
The investigators will conduct an observational study comparing the number of bleeding days before and after contraceptive implant (Nexplanon) replacement.

DETAILED DESCRIPTION:
There is very limited information regarding number of bleeding days after replacement of the contraceptive implants (Nexplanon). More detailed information on this topic will help clinicians counsel patients and help women decide if they would like to pursue contraceptive implant replacement.

The investigators will conduct a prospective cohort study of (N=114) among women replacing their contraceptive implant. The primary outcome of the study is the difference in number of bleeding days between the 4-week periods before and after implant replacement. Secondary outcomes include satisfaction with bleeding. Additionally, a secondary outcome will be the number of bleeding days in month 2 and month 3 after replacement of the contraceptive implant. The outcomes will be measured in bleeding diaries and satisfaction surveys.

Through a text messaging application, the investigators will send the participants hyperlinks to the diaries/surveys at the stated time points. Participants will report if they had bleeding and the amount based on the Pictorial Blood Assessment Chart (Higham). Participants will complete weekly surveys regarding their satisfaction with their bleeding utilizing a Likert scale. The investigators will also ask participants to complete a survey regarding their satisfaction with their bleeding at end of month 2 and at the end of month 3 after replacement of their contraceptive implant.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women 18-50 years old
* With a contraceptive implant (for patient participants)
* Able to consent in English
* Palpable contraceptive implant

Exclusion Criteria:

* Non-palpable contraceptive implant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients scheduled at UC San Diego for a contraceptive implant after approximately 3 years (32-40 months) of use.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of bleeding days during 4 weeks before replacement | 4 weeks (28 days) before day of implant replacement.
  Number of days participants experienced bleeding during the 4 weeks before implant replacement.
Number of bleeding days 4 weeks after replacement | 4 weeks (28 days) after day of implant replacement
  Number of days participants experienced bleeding during the 4 weeks after implant replacement.

SECONDARY OUTCOMES:
Satisfaction with bleeding before replacement | 4 weeks (28 days) before day of implant replacement
  Using a 1-5 Likert scale with 1=Not Satisfied and 5=Very Satisfied, participants will report satisfaction with their bleeding before implant replacement.
Satisfaction with bleeding after replacement | 4 weeks (28 days) after day of implant replacement
  Using a 1-5 Likert scale with 1=Not Satisfied and 5=Very Satisfied, participants will report satisfaction with their bleeding after replacement
Number of bleeding days during the second month after implant replacement | Second month (defined as 29-56 days) after implant replacement
  Number of days participants experienced bleeding during the second month after implant replacement
Number of bleeding days during the third month post replacement | Third month (defined as 57-84 days) after implant replacement
  Number of days participants experienced bleeding during the third month after implant replacement

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Higham JM, O'Brien PM, Shaw RW. Assessment of menstrual blood loss using a pictorial chart. Br J Obstet Gynaecol. 1990 Aug;97(8):734-9. doi: 10.1111/j.1471-0528.1990.tb16249.x. PMID 2400752